CLINICAL TRIAL: NCT06850493
Title: The Impact of a Preoperative Very Low Calorie Ketogenic Diet (VLCKD) on Body Composition in Patients Undergoing Bariatric Surgery: a Randomised Controlled Trial
Brief Title: Ketogenic Diet Prior to Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Aliyar Esfandiyari Noushi, Doctor of Medicine, Maxima Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL81550.015.22
Record Dates: First submitted 2024-07-30; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery Candidate; Ketogenic Dieting
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VLCD (Very-Low-Calorie-Diet) (Active Comparator): Patients in the VLCD group receive, as prescribed by a dietician, three meal sachets a day.
  Each meal contains ±240kcal (=1004 kJ), 17-20g carbohydrates and 14-17g proteins.
  Altogether, this diet contains less than 800 kcal/day, 50-60g carbohydrates per day and 42-51g protein per day. The diet is continued for 14 days, until the day prior to surgery. In addition to using liquid meals, patients are allowed to consume raw vegetables (e.g., endive, spinach, cucumber, lettuce; without oil or dressings), and clear soups. Patients are advised to drink at least two liters per day of mineral water, tea, infusions or coffee without milk and/or sugar.
  Interventions: Dietary Supplement: VLCD (Very-low-calorie-diet)
- VLCKD (Very-Low-Calorie-Ketogenic-Diet) (Active Comparator): Six meal sachets are given to patients in the VLCKD group each day. A single meal has 16-19g of proteins, 2-3g of carbohydrates, and ±86kcal (=363 kJ). Together, the daily energy intake from this diet is less than 800 kcal, 50 g of carbohydrates, and 100 g of proteins. The diet is followed up to the day before surgery for a total of 14 days. Patients are recommended to ingest vegetables with a low glycaemic load (such as sprouts, lettuce, spinach, and tomatoes) in addition to the liquid meals. Patients are encouraged to consume at least two liters of mineral water, tea, infusions, or coffee without milk or sugar each day.
  Interventions: Dietary Supplement: VLCKD (ketogenic diet)

INTERVENTIONS:
Dietary Supplement: VLCKD (ketogenic diet) — diets prior to bariatric surgery
  Other Names: VLCKD
  Arms: VLCKD (Very-Low-Calorie-Ketogenic-Diet)
Dietary Supplement: VLCD (Very-low-calorie-diet) — diets prior to bariatric surgery
  Other Names: VLCD
  Arms: VLCD (Very-Low-Calorie-Diet)

SUMMARY:
Standard dietary regiments for bariatric are advised prior to surgery. The most used diet is a very low calorie diet (VLCD). These diets potentially have multiple pittfalls.

Very low-calorie ketogenic diets (VLCKD) have been proposed as a new regimen for achieving weight- and liver volume loss in patients undergoing bariatric surgery. The beneficial effect of VLCKDs compared to (V)LCDs is the aimed preservation of FFM and RMR, while still reducing FM. Only a few small studies addressed the role of VLCKDs prior to bariatric surgery, and the data including FFM and FM is actually scarce. Therefore, a well-designed randomised controlled trial is necessary to establish the efficacy of a VLCKD.

DETAILED DESCRIPTION:
According to the World Health Organization, obesity rates have nearly tripled since 1975, resulting in the mortality of four million individuals each year. Obesity contributes to a reduced quality of life and is a significant risk factor for multiple chronic diseases such as type 2 diabetes mellitus, cardiovascular disease, osteoarthritis and certain types of cancer . Bariatric surgery is regarded the most effective treatment for extreme obesity because it achieves significant long-term weight loss and improves or even eliminates obesity-related complications. Based on the American Society for Metabolic and Bariatric surgery, approximately 230.000 bariatric procedures are performed annually, and those procedures predominantly included sleeve gastrectomy and Roux-en-Y gastric bypass (RYGB) procedures. Bariatric surgery can be challenging because of an increased thickness of the abdominal wall, the presence of intra-abdominal obesity and hepatomegaly. These anatomical changes are associated with more anaesthetic and surgical manoeuvres during the procedure. Losing weight prior to the procedure is frequently advised because it may help to overcome technical challenges. It may furthermore improve short-term outcomes like surgical time, blood loss, hospital stay and postoperative complications, as well as long-term outcomes like weight loss.

In the preoperative phase, weight loss can be realised by multiple dietary regimens, including low-calorie diets (LCD) (800-1500 kcal/day) and very low-calorie diets (VLCD) (<800 kcal/day). In Máxima Medical Center and a few other hospitals performing bariatric surgery in the Netherlands, the VLCD is the standard diet of choice, which begins two weeks prior to surgery. Systematic reviews reported, as result of these diets, a reduction in liver size (5-20% with a VLCD; 12-27% with a LCD), intrahepatic fat (43% with a VLCD; 40-51% with a LCD) and body weight (2.8-14.8kg with a VLCD; 5.4-23.6kg with a LCD). These diets varied in duration, from two weeks to four months. One of the primary drawbacks of these diets is the loss of metabolically active fat free mass (FFM) and lean body mass (LBM), which are crucial for whole-body protein metabolism, in addition to fat mass (FM). In contrast to FFM, LBM contains bone mass, connective tissue, internal organs and essential fat stored in these tissues. It has been hypothesised that LBM will contain 3 to 5% more fat than FFM. A significant loss of FFM may negatively affect the resting metabolic rate (RMR), slow the rate of weight loss and predispose weight regain in the long-term. A significant loss of FFM, in continuing presence of an excessive FM, may furthermore contribute to sarcopenic obesity. A second important downfall is that some patients may not tolerate a (V)LCD regime due to side-effects leading to poor compliance and subsequently poor weight loss outcomes. For clinical trials, the reported attrition rate for a (V)LCD regime is around 20%, raising concerns about the study validity.

Very low-calorie ketogenic diets (VLCKD) have been proposed as a new regimen for achieving weight- and liver volume loss in patients undergoing bariatric surgery. A VLCKD is characterized by a very low carbohydrate content (<50 g/daily), a low-fat content (15-30 g fat/daily) and a high amount of proteins (1-1.5 g protein/kg ideal body weight). The beneficial effect of VLCKDs compared to (V)LCDs is the aimed preservation of FFM and RMR, while still reducing FM. In addition, the compliance of patients might be improved by VLCKDs, possibly due to the anorexigenic effect and hunger reduction of ketone bodies. Only a few small studies addressed the role of VLCKDs prior to bariatric surgery, and the data including FFM and FM is actually scarce. A retrospective cohort study found that a three-week lasting VLCKD resulted in more weight loss (5.8kg vs. 4.8kg) compared to a VLCD. In addition, two prospective cohort studies showed as result of a VLCKD, FFM was reduced by 7.6 kg (10.0%) and 0.7kg (1.1%) , whereas FM was reduced by 10.5kg (17.9%) and 5kg (8.8%). What is important to note is that these studies lack a control group, randomisation and are subjected to limitations in FFM and FM measurement due to the use of single-frequency bioelectrical impedance analysis (BIA). Therefore, a well-designed randomised controlled trial is necessary to establish the efficacy of a VLCKD.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for bariatric surgery (≥35 kg/m2 with obesity-related comorbidities, or a BMI of

  * 40 kg/m2 with or without comorbidities)
* Roux-en-Y Gastric bypass (RYGB)

Exclusion Criteria:

* Weighing over 150kg because this amount is a limitation by the DXA device
* Diabetes mellitus type 1
* Allergic to milk proteins
* A recent history of a heart attack (< 12 months), heart failure or cardiac arrhythmias
* Kidney and/or liver failure (creatinine levels >1.3 mg/dl or liver enzyme levels (AST, ALT, GGT)) less than three times over the upper normal threshold
* Current infectious, sepsis or malignant disease
* Rare condition like galactosemia, phenylketonuria or porphyria
* Persistent diarrhoea
* Hypokalaemia, chronic therapies with diuretics as furosemide and hydrochlorothiazide
* Pregnancy or plans to get pregnant in the coming months
* Patients who did not meet criteria to be eligible for bariatric surgery (BMI <35, psychological or unstable psychiatric disorders, inadequate dietary regimen or inadequate exercise pattern which can't be resolved in the upcoming 6 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in FFM (%) in proportion to TBWL | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  The main outcomes are the change in FFM (percentage) in proportion to total body weight loss (TBWL) measured from baseline to two weeks after start of the diet.

SECONDARY OUTCOMES:
Change in weight | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Weight (in kilograms), measured by Multi-frequency bioelectrical impedance analysis (MF-BIA), measured a total of three times. Twice before surgery: once prior to the diet and once after ending the diet. The last time 3 months after surgery
Physical activity questionnaire | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Measured by International Physical Activity Questionnaire (IPAQ). The IPAQ is used to estimate physical activity levels and to examine if there are differences in comparison to each diet and to assess differences preoperatively and postoperatively during and after completion of the diet.
  Measured in minutes per day. With a minimum of 0 minutes up to 1440 minutes a day.
  Higher scores might indicate higher levels of activity
Patient satisfaction assessed by a questionnaire | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  5-point Likert scale: not at all satisfied, slightly satisfied, neutral, very satisfied and extremely satisfied). To assess the degree of contentment in regard to each diet. Higher scores results in more satisfaction
Incidence of side effects, assesed by questionnaire | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Measured by self-reported questionnaires, making use of a dichotomous scale (Yes; No).
  With a score Yes indicating the occurence of a side effect.
Compliance assesed by return of diet sachets | 2 weeks prior to surgery till the day of surgery
  Via the amount of sachets a patient has used. The patients has to bring the empty sachets along to their appointment. With the amount of sachets we will have insight to how many have been used and to the extent of compliance a patient has shown regarding their dietary intake. More sachets returned mean a possibly a higher compliance
Change in weight | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Weight (in kilograms), measured by and Dual energy x-ray absorptiometry (DXA), measured twice before surgery (prior to the diet and after ending the diet) and once three months after surgery.
Upper extremity muscle strenght | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Muscle strength (in kilogram), measured by handgrip peak strength, measured twice before surgery (prior to start diet and after finishing diet) and measured after surgery. Muscle strength is tested to map general upper extremity muscle strength.
Surgical outcome (1) | Day of surgery
  Surgical time needed to perform the RYGB. Measured in minutes
Surgical outcome (2) | From day of surgery untill the day of discharge, counted as the nights a patient has stayed in the hospital for admission
  Hospital stay during admission. Measured in days.
Surgical outcome (3) | Day of surgery up to 30 days postoperatively
  Complications occuring during admission up to 30 days postoperatively. Scored with a yes or no
Surgical outcome (4) | Day of surgery up to 30 days postoperatively
  Re-admissions occuring within 30 days postoperatively. Scored with yes or no
Biochemical testing- Ketosis | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  B-hydroxybutyrate measurement in blood. Aim of this test is to measure the degree of ketosis. Elevated levels of B-hydroxybutyrate could indicate a state of ketosis
Biochemical testing (Electrolytes- Sodium) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Sodium. Reference values between 135-145 mmol/L are seen as normal. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Electrolytes - Potassium) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Potassium. Reference values of 3.5-5.0 mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Electrolytes - Albumin) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Albumin. Reference values of 31-44g/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Liverfunction - Aspartate Aminotransferase (AST)) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Aspartate Aminotransferase (AST). Reference values of <31 U/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Liverfunction - Alanine Transaminase (ALT)) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Alanine Transaminase (ALT). Referene values of <34 U/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Liverfunction - Gamma glutamyl transpeptidase (GGT)) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Gamma glutamyl transpeptidase (GGT). Reference values of <38 U/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Kidney function - Creatinine) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Creatinine. Reference values of 49-90 micromol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Kidney function - Urea) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Urea. Reference values of 2.5-6.4 mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Kidney Function - Estimated glomerular filtration rate (eGFR)) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Estimated glomerular filtration rate (eGFR). Reference values of >90 ml/min/1.73m2. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Iron) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Iron. Reference values of 9-30 micromol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Hemoglobin) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Hemoglobin. Reference values ranging from 7.5-10 mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Metabolic profile - Total cholesterol) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Total cholesterol. Reference value < 5mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Metabolic profile - low-density lipoprotein (LDL)) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Low-density lipoprotein (LDL). Reference value <2.6mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Metabolic profile - High-density lipoprotein (HDL)) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  High-density lipoprotein (HDL). Reference value >1.1 mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Metabolic profile - Triglycerides) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Triglycerides. Reference value <2.0 mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Calcium) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Calcium. Reference values ranging from 2.10-2.55 mmol/L. Aim of the biochemical testing is to assess nutritional status
Biochemical testing (Glucose) | 2 weeks prior to surgery, day of surgery and 3 months after surgery
  Glucose. Reference values ranging from 4.0-7.8 mmol/L. Aim of the biochemical testing is to assess nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Francois van Dielen, MD PhD, Principal Investigator — Maxima Medical Center
Locations (1):
- Maxima Medical Center, Veldhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No